CLINICAL TRIAL: NCT03601624
Title: Multicenter Study of Pomalidomide, Cyclophosphamide, and Dexamethasone in Relapsed Refractory Myeloma: Safety Profile in Mexican Population
Brief Title: Pomalidomide/Cyclophosphamide/Dexamethasone in Relapse Refractory Myeloma: Safety Profile in Mexicans
Acronym: MM-POM-2018
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Martha Alvarado Ibarra, Chief of Hematology Area, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSSTE-POM-CY-MM-2018
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma Progression; Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Relapse; Progression; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Disease Progression | interventions — pomalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Interventional phase 2, multicentric, open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 1. Pomalidomide at 4 mg orally on days 1-21 of a 28 day cycle
  2. Cyclophosphamide 300 mg IV on days 1 and 15 of a 28 day cycle.
  3. Dexamethasone 40 mg PO weekly.(Or 20 mg if patients are older than 75 years )
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — 1. Pomalidomide at 4 mg orally on days 1-21 of a 28 day cycle
  2. Cyclophosphamide 300 mg IV on days 1 and 15 of a 28 day cycle.
  3. Dexamethasone 40 mg PO weekly.(Or 20 mg if patients are older than 75 years )
  Other Names: Cyclophosphamide; Dexamethasone

SUMMARY:
Despite available therapies, MM uniformly fatal and participants who have received prior lenalidomide (Len) and bortezomib have a median overall survival (OS) of 9 months.

Pomalidomide (Pom) plus low-dose dexamethasone (Dex) significantly improved efficacy parameters in terms of progression free survival (PFS), OS, and overall response (ORR) compared with high-dose Dex in participants with refractory or relapsed, and refractory MM, including participants with disease refractory to both bortezomib and lenalidomide.

Alkylating agents also represent standard therapies for participants with MM. There are some reports demonstrating combination of Len and continuous cyclophosphamide (Cy) achieve an ORR of 50% in Len refractory participants, suggesting Cy may be able to overcome resistance to Len.

The investigators aimed to assess the safety in Mexican MM participants in relapse/refractory stage of the triple combination: IV Cy in combination with Pom plus Dex until disease progression. A multicenter study is proposed.

Primary endpoint: Safety. Efficacy as secondary endpoint: PF, OS and ORR.

DETAILED DESCRIPTION:
Multiple myeloma is a plasma cell malignancy with accounts for about 1% of all cancers. Despite available therapies, the disease remains uniformly fatal and participants who have received prior lenalidomide and bortezomib have a median overall survival of 9 months.

Combination therapy is often used in clinical practice. In an attempt to overcome drug/clone resistance, other report with pomalidomide, dexamethasone and cyclophosphamide (PomCyDex) show efficacy and safety information, regimen for refractory myeloma patients with higher overall response rate than pomalidomide and dexamethasone.

In this case a phase II trial scheme is proposed: 1. Pomalidomide at 4 mg orally on days 1-21 of a 28 day cycle, 2. Cyclophosphamide 300 mg IV on days 1 and 15 of a 28 day cycle; and 3. Dexamethasone 40 mg PO weekly. Participants who were >75 years of age or those who were known to be intolerant to 40 mg weekly dexamethasone are going to receive 20 mg dexamethasone on the same schedule.

Pomalidomide is a drug wide studied in American and European population, but not in México. Even it has been approved by local Regulatory authority, there is not any trial supporting data about safety and efficacy in Mexican population. Alkylating agents are very active in MM, and in combination with novel therapies, such as immunomodulatory drugs, has shown to enhance efficacy in relapsed/refractory setting.

It is proposed phase 2 study to assess safety and efficacy of treatment with Pomalidomide in combination with Cyclophosphamide and dexamethasone in a sample of Mexican RRMM participants from ISSSTE.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old
2. Relapsed and refractory multiple myeloma patients that had received ≥2 prior lines of therapies including a proteasome inhibitor and Lenalidomide; if cyclophosphamide was included in a previous line, complete scheme has to be finished at least 6 months previously to initiate in this IIT.
3. Measurable disease as defined by the presence of 1 of the following: serum monoclonal protein ≥0.5 g/dL; urine monoclonal protein >200 mg/24 h; or serum involved free light chain ≥10 mg/dL and abnormal serum free light chain ratio.
4. ECOG 0 to 2
5. Serum creatinine level <3mg/dL.
6. Absolute neutrophil count ≥1000/mm3, and a platelet count ≥30 000/mm3.
7. Females of childbearing potential has to have a negative serum or urine pregnancy test within 10 to 14 days prior to, and within 24 hours of, starting pomalidomide.
8. A washout period of 2 weeks prior to cycle 1 day 1 from prior therapies are required.

Exclusion Criteria:

1. Patients with known hypersensitivity to thalidomide or lenalidomide
2. Patients who had HIV or active hepatitis B or C;
3. Patients with grade 3 or more neuropathy
4. Patients with active malignancy requiring therapy within the next year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of Treatment - Emergent Adverse Events | 2 years
  Adverse events leading to death or to discontinuation from treatment, events classified grade 3 or higher, study drug-related events, and serious adverse events are going to be listed separately.

SECONDARY OUTCOMES:
Efficacy as secondary endpoints: progression free survival, overall survival and overall response rate | 2 years
  For the secondary end point, ORR and its 95% confidence interval are going to be calculated for the study groups using the exact binomial method

CONTACTS AND LOCATIONS:
Overall Officials: MARTHA ALVARADO, MD, Principal Investigator — Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Locations (1):
- ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richardson PG, Mark TM, Lacy MQ. Pomalidomide: new immunomodulatory agent with potent antiproliferative effects. Crit Rev Oncol Hematol. 2013 Oct;88 Suppl 1:S36-44. doi: 10.1016/j.critrevonc.2013.02.001. Epub 2013 Jun 17. PMID 23786844
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Dimopoulos MA, Leleu X, Palumbo A, Moreau P, Delforge M, Cavo M, Ludwig H, Morgan GJ, Davies FE, Sonneveld P, Schey SA, Zweegman S, Hansson M, Weisel K, Mateos MV, Facon T, Miguel JF. Expert panel consensus statement on the optimal use of pomalidomide in relapsed and refractory multiple myeloma. Leukemia. 2014 Aug;28(8):1573-85. doi: 10.1038/leu.2014.60. Epub 2014 Feb 5. PMID 24496300
- [Background] Baz RC, Martin TG 3rd, Lin HY, Zhao X, Shain KH, Cho HJ, Wolf JL, Mahindra A, Chari A, Sullivan DM, Nardelli LA, Lau K, Alsina M, Jagannath S. Randomized multicenter phase 2 study of pomalidomide, cyclophosphamide, and dexamethasone in relapsed refractory myeloma. Blood. 2016 May 26;127(21):2561-8. doi: 10.1182/blood-2015-11-682518. Epub 2016 Mar 1. PMID 26932802
- [Background] Martha Alvarado Ibarra, Manuel López Hernández, José LuisAlvarez Vera, Maricela Ortiz Zepeda, Verónica Mena Zepeda and Eugenia Espitia Ríos. Outcomes and Evolution In The Tratment Of Multiple Myeloma In The Last 20 Years Experience Of A Mexican Institution. International Journal of Information Research and Review 3(9):2811-2817, 2016